CLINICAL TRIAL: NCT05114577
Title: Recovery Sleepers: A Pilot Study of a Sleep Health Intervention for College Students in Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Society for Health Psychology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HM20022646
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Sleep; Addiction
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery Sleepers program. (Experimental)
  Interventions: Behavioral: Recovery Sleepers program.
- Email recommendations (Placebo Comparator)
  Interventions: Behavioral: Email recommendations

INTERVENTIONS:
Behavioral: Recovery Sleepers program. — Attend two, 90-minute remote discussion groups (~10 other participants and 2 study team members) via Zoom. During these groups, participants will receive educational materials about how to improve sleep. They will also discuss sleep and sleep-related behaviors, including how active substance use and recovery may have changed sleep, with a small group of other participants.
  Arms: Recovery Sleepers program.
Behavioral: Email recommendations — Receive recommendations (via email) to help improve sleep
  Arms: Email recommendations

SUMMARY:
The purpose of this research study is to examine how to improve sleep in college students in recovery from substance use disorder(s). This study is a pilot test of an experimental program called Recovery Sleepers (RS) to explore its feasibility and how well it works to improve sleep, wellbeing, and cravings.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age
* Enrolled (full- or part-time) at a college or university
* Have struggled with substance addiction in the past
* More than 3 months of self-reported continuous abstinence from alcohol and all illegal drugs
* Have an Internet-enabled device with audio capabilities.

Exclusion Criteria:

* Younger than 18 years of age
* Not enrolled at VCU
* Have not struggled with substance addiction in the past
* Have not had at least 3 months of self-reported continuous abstinence from alcohol and all
* illegal drugs
* In active treatment for a sleep disorder (seen a health provider specifically regarding sleep within the last 6 months)
* Unable to communicate in English both orally and in writing
* Do not have an Internet-enabled device with audio capabilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-24 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Satisfaction with treatment | 6 weeks
  Participants will rate their experiences in the study using a scale from 1 (Strongly disagree) to 5 (Strongly agree). Treatment and placebo groups will answer a different number of questions. Scores will be averaged to yield a single score between 1 and 5.
Study participant retention | 6 weeks
  Percent of participants who complete all 6 weeks of the study
Study material completion | 6 weeks
  Percent of participant who complete all of the study materials over the course of the study
Study group attendance | 6 weeks
  Percent of participants who attend all study group meetings
Recruitment success | Baseline
  Number of participants recruited into the study

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Dautovich, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No